CLINICAL TRIAL: NCT06856681
Title: A Study of the Clinical Effect of the Implementation of a Blood Biomarker Into Memory Clinics in the Department of Veterans Affairs and Other Closed System Healthcare Memory and Dementia Sites in the United States
Brief Title: Clinical Utility of Early vs. Late Blood Biomarker Testing for Alzheimer's Disease
Acronym: ADELAIDE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor decision to cancel project before enrollment.
Sponsor: C2N Diagnostics (Industry)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 250
Record Dates: First submitted 2025-02-06; First posted 2025-03-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Alzheimers Disease
Keywords: Blood biomarkers; Mild Cognitive Impairment; Dementia; Alzheimers disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment interventional model in which participants are randomized into one of two groups to evaluate the impact of the timing of PrecivityAD2 test on physician diagnostic confidence and clinical decision-making. Participants in the early testing group receive their PrecivityAD2 test at Visit 1, while those in the delayed testing group receive their results at Visit 3 (Day 90). Both groups proceed independently through the study, and assessments occur at standardized time points to measure changes in diagnostic confidence, treatment decision, and diagnostic test utilization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Testing Group (Cohort A) (Experimental): Participants in this group will have blood drawn from the PrecivityAD2 test at Visit 1 (Day 0). Physicians will use these results in clinical decision-making from that point forward.
  Interventions: Diagnostic Test: PrecivityAD2 - Early Testing
- Delayed Testing Group (Cohort B) (Experimental): Participants in this group will have blood drawn for the PrecivityAD2 test at Visit 2 (Day 90). Until then, standard clinical decision-making will process without access to PrecivityAD2 results.
  Interventions: Diagnostic Test: PrecivityAD2 - Delayed Testing

INTERVENTIONS:
Diagnostic Test: PrecivityAD2 - Early Testing — Participants in Cohort A will receive PrecivityAD2 testing at Visit 1, with results disclosed shortly after testing.
  Arms: Early Testing Group (Cohort A)
Diagnostic Test: PrecivityAD2 - Delayed Testing — Participants in Cohort B will receive PrecivityAD2 testing at Visit 2, with results disclosed shortly after testing.
  Arms: Delayed Testing Group (Cohort B)

SUMMARY:
The goal of this study is to evaluate whether use of the PrecivityAD2 blood biomarker assay with early result disclosure along with discretionary Precivity-ApoE proteotype testing will shorten the time to Alzheimer's Disease or non-Alzheimer's diagnosis as compared to delayed result disclosure.

Participants will be randomized into the early PrecivityAD2 blood biomarker test & disclosure group (Cohort A) or to the later PrecivityAD2 blood biomarker test & disclosure group (Cohort B) where blood samples will be collected and tested using the PrecivityAD2 test at Visit 1 (day 0) and Visit 2 (day 90). Participants will attend study visits for one year after their enrollment. An optional sub-study will be offered to collect information through questionnaires at each visit regarding participant's and their care-giver's experiences through the AD diagnostic journey.

DETAILED DESCRIPTION:
Healthcare providers engaged in memory care and Alzheimer's disease (AD) management have shown significant interest in the performance of plasma tests. A collaboration with Veteran's Affairs (VA) and other closed healthcare systems represents an opportunity to examine the clinical validity and utility of blood biomarkers (BBM). The ADELAIDE study is a prospective, randomized, clinical utility, economic impact and real-world study. The BBM test under study is the PrecivityAD2 blood test that uses high-resolution liquid chromatography mass spectrometry to measure plasma Aβ42/40 and p-tau217/np-tau217 ratios. This study will assess and quantify the impact of BBM testing to overall time-to-diagnosis and time to prescription of an appropriate Alzheimer's Disease (AD) or non-AD therapy. Additionally, this study will assess the impact of BBM testing to procedure utilization and overall costs of healthcare and will assess the diagnostic confidence of clinicians that order the test.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age: 50 years.
2. Patients presenting with symptoms of mild cognitive impairment (MCI) or other cognitive impairments in which the enrolling clinician clinically suspects Alzheimer's pathology as the primary cause of symptomatic presentation
3. Patients presenting with mixed brain pathologies including MCI/ cognitive impairments in which the investigator clinically suspects Alzheimer's pathology as the primary or contributing cause of symptomatic presentation
4. Patients are able to attend study visits and standard care visits over the period of 1 year from the date of enrollment
5. Patients are able to undergo routine phlebotomy and provide up to six (6) 10 ml tube(s) of blood for study related tests plus any additional blood necessary for standard laboratory testing at each study timepoint
6. Patients are able to undergo standard care diagnostic procedures to include MRI (or CT), amyloid PET and/or CSF biomarker testing for AD diagnosis if prescribed by investigator
7. Patients are able to provide informed consent. Or, if in the opinion of the clinician, the patient is unable to adequately understand the nature of the trial and protocol requirements, a family member or appropriate representative of the patient is present to consent, with additional assent by the patient.

Exclusion Criteria

1. Patients younger than 50 years of age
2. Patients being evaluated for cognitive impairment known to be predominantly the result of a disease or condition other than AD
3. Patients previously diagnosed with AD, unless the ADELAIDE investigator has a strong clinical suspicion suggestive of an incorrect initial diagnosis upon referral
4. Patients with no cognitive impairment or clinical symptoms of AD
5. Patients desiring genetic testing for Alzheimer's disease markers without current cognitive impairment or other relevant clinical symptoms
6. Patients who are not able or not willing to undergo standard care diagnostic procedures to include MRI (or CT), amyloid PET and/or CSF biomarker testing for AD diagnosis as prescribed by investigator
7. Patients who are not able to understand the nature of the study nor the study requirements and not represented by a family member or other appropriate representative who is able to consent on behalf of the patient
8. Patients who are not able to commit to attending the required study and/or standard care visits
9. Patients who are not able to undergo routine phlebotomy or provide blood samples in the quantity required by the study protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Time to achieve >=90% Diagnostic Confidence for AD or Non-AD | From enrollment until diagnosis, with primary assessment at Visit 2 (Day 90) and Visit 3 (Day 180).
  Number of days from enrollment to achieving a diagnostic confidence score of >=90% for AD or non-AD diagnosis (based on physician survey).
Proportion of Patients with AD of Non-AD Diagnosis | Assessed at Visit 2 (Day 90) and Visit 3 (Day 180)
  Proportion of patients with a confirmed AD or non-AD diagnosis with a diagnostic confidence score of >=90%.

SECONDARY OUTCOMES:
Time to Initiation or Modification of AD or Non-AD Therapy | Measured from enrollment through Visit 4 (Day 365).
  Number of days from enrollment to the prescription, initiation, or modification of an AD or non-AD therapy. Data will be sourced from medical records and recorded in eCRF.
Proportion of patients on AD or non-AD prescription | Assessed at Visit 3 (150-210)
  Proportion of patients on AD or non-AD prescription (e.g., DMT, treatments for DLB/PDD or VaD, cholinesterase inhibitors, other) at Visit 3 (150-210).
Number and Type of Diagnostic Tests Ordered | Evaluated cumulatively at Visit 2 (Day 90), Visit 3 (Day 180), and Visit 4 (Day 365)
  Total number and type of additional diagnostic tests ordered (e.g., amyloid PET, MRI, CSF biomarkers) from Visit 2 (Day 90) through the date of AD or non-AD diagnosis with physician confidence >=90%. Data will be collected via physician-reported case forms.
Change in Physician Diagnostic Confidence | Collected at Enrollment/Baseline (Day 0), Visit 2 (Day 90), Visit 3 (Day 180) and Visit 4 (Day 365)
  Comparison of physician reported confidence of AD or non-AD diagnosis (0-100%) before and after receiving PrecivityAD2 results. Confidence scores will be collected by physician survey.

OTHER OUTCOMES:
Patient-Reported Experience with Diagnostic Process | Collected at Visit 2 (Day 90), Visit 3 (Day 180) and Visit 4 (Day 365)
  Patient-reported experience with the diagnostic journey, including perception of the clarity and utility of PrecivityAD2 results. Assessed using patient surveys.
Caregiver-Reported Perception of Disease Burden | Collected at Visit 2 (Day 90), Visit 3 (Day 180) and Visit 4 (Day 365)
  Caregiver-reported assessment of disease burden, changes in the patient's condition, and perceived impact on daily life. Collected through structured caregiver surveys.
Healthcare Utilization and Costs | Enrollment through Visit 4 (Day 365)
  Total healthcare costs associated with diagnostic evaluations, physician visits, and treatments. Healthcare utilization and cost data will be collected from medical records and analyzed retrospectively after Visit 4 (Day 365).

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Neurology, Study Director — C2N Diagnostics

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meyer MR, Kirmess KM, Eastwood S, Wente-Roth TL, Irvin F, Holubasch MS, Venkatesh V, Fogelman I, Monane M, Hanna L, Rabinovici GD, Siegel BA, Whitmer RA, Apgar C, Bateman RJ, Holtzman DM, Irizarry M, Verbel D, Sachdev P, Ito S, Contois J, Yarasheski KE, Braunstein JB, Verghese PB, West T. Clinical validation of the PrecivityAD2 blood test: A mass spectrometry-based test with algorithm combining %p-tau217 and Abeta42/40 ratio to identify presence of brain amyloid. Alzheimers Dement. 2024 May;20(5):3179-3192. doi: 10.1002/alz.13764. Epub 2024 Mar 16. PMID 38491912
- [Background] Palmqvist S, Tideman P, Mattsson-Carlgren N, Schindler SE, Smith R, Ossenkoppele R, Calling S, West T, Monane M, Verghese PB, Braunstein JB, Blennow K, Janelidze S, Stomrud E, Salvado G, Hansson O. Blood Biomarkers to Detect Alzheimer Disease in Primary Care and Secondary Care. JAMA. 2024 Oct 15;332(15):1245-1257. doi: 10.1001/jama.2024.13855. PMID 39068545
- [Background] Schindler SE, Galasko D, Pereira AC, Rabinovici GD, Salloway S, Suarez-Calvet M, Khachaturian AS, Mielke MM, Udeh-Momoh C, Weiss J, Batrla R, Bozeat S, Dwyer JR, Holzapfel D, Jones DR, Murray JF, Partrick KA, Scholler E, Vradenburg G, Young D, Algeciras-Schimnich A, Aubrecht J, Braunstein JB, Hendrix J, Hu YH, Mattke S, Monane M, Reilly D, Somers E, Teunissen CE, Shobin E, Vanderstichele H, Weiner MW, Wilson D, Hansson O. Acceptable performance of blood biomarker tests of amyloid pathology - recommendations from the Global CEO Initiative on Alzheimer's Disease. Nat Rev Neurol. 2024 Jul;20(7):426-439. doi: 10.1038/s41582-024-00977-5. Epub 2024 Jun 12. PMID 38866966